CLINICAL TRIAL: NCT04982809
Title: Effectiveness and Pharmacoeconomic Study of Using Different Corticosteroids in the Treatment of Interstitial Lung Diseases
Brief Title: Cost-effectiveness Analysis of Three Corticosteroids in ILDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa G. Elhennawy, Assistant Lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (2183)
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Betamethasone; Dexamethasone; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Betamethasone group (Active Comparator)
  Interventions: Drug: Betamethasone, Dexamethasone, Prednisolone
- Dexamethasone group (Active Comparator)
  Interventions: Drug: Betamethasone, Dexamethasone, Prednisolone
- Prednisolone group (Active Comparator)
  Interventions: Drug: Betamethasone, Dexamethasone, Prednisolone

INTERVENTIONS:
Drug: Betamethasone, Dexamethasone, Prednisolone — Corticosteroids

SUMMARY:
This was a 3 months prospective, open label, and parallel study to test the efficacy of 3 different corticosteroids in the management of interstitial lung diseases. Followed by a pharmacoeconomic analysis to find which regimen (betamethasone, dexamethasone or prednisolone) is the most cost-effective.

DETAILED DESCRIPTION:
Three different corticosteroid regimens were evaluated for the management of interstitial lung diseases (ILDs) with specific focus on hypersensitivity pneumonitis (HP) where the patients were divided into 3 treatment groups:

* Group I: patients receiving weekly pulse doses of betamethasone IM injection (equivalent dose to that of prednisolone daily dose in a week).
* Group II: patients receiving weekly pulse doses of dexamethasone IV injection (equivalent dose to that of prednisolone daily dose in a week).
* Group III: patients receiving oral prednisolone daily (dose range 15-20 mg/day).

  10 mg oral prednisolone oral ≡ 1.5 mg dexamethasone intravenous ≡ 1.2 mg betamethasone intramuscular.

After the administration of the above-mentioned medications, the patients were followed-up over 3 months to evaluate their disease progression. Informed consent was obtained from all subjects or their surrogate after explanation and understanding of the nature, purpose, and potential risks of the study. The study protocol was approved by the Ethics Committee, Faculty of Pharmacy, Cairo University (protocol serial number: CL (2183)) .

A special patient information sheet was designed to collect all information required for data analysis. The sheet was designed to be divided into several sections:

1. Demographic Data The first section of the patients' information sheet was designed to accommodate the basic general and demographic data (name, address, age, telephone number, social status, weight, and height of the patient). These details were documented from the patient's medical notes.
2. Medical Data Medical records were used to obtain other data including date and time of examination, the diagnosis, medications on recruitment (if any), smoking habits, patient's medical history, in addition to the patient's medication history.
3. Parameters Used to Measure Effectiveness as KL-6, PFTs, ESR, CRP
4. Parameters to Evaluate Treatment Safety Liver Function Tests, Random Blood Glucose (RBG), Blood Pressure

Cost Effectiveness Analysis The study is designed from patient perspective where the direct medical costs as well as the indirect costs (e.g., loss of patients' income) are studied. The costs are collected directly from the patient prospectively throughout the study period. All costs were actual covering the treatment expenses as: the cost of the medications, the cost of administration, the cost of the hospital stay due to ILD during the study period, the cost of the physician's visit and the cost afforded by the patient in order to administer the recommended medication, any extra costs due to exacerbations or adverse effects due to the use of corticosteroids and costs of transportation and days-off.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ILD (hypersensitivity pneumonitis) with age between18 and 65 years old.
* Symptoms including dry cough and shortness of breath.
* Significant decrease in pulmonary function (desaturation by 4% after 6-minute walk distance), where the patients were no more controlled on their prednisolone maintenance therapy (up to 10 mg/day).
* Chest CT showing ground glass opacity and band of shadow.

Exclusion Criteria:

* Patients with any other organ affliction (heart failure (ejection fraction 40-50%), renal failure (decrease in glomerular filtration rate > 75%), or liver cirrhosis (transient elastography liver stiffness measurements 12.5-75.5 kPa)).
* Active infection.
* Patients on other immunosuppressive medications (e.g., cyclophosphamide) and anti-fibrotic (e.g., interferon, pirfenidone, endothelin-1 antagonist and tumor necrosis factor α modulator).
* History of pulmonary embolism (corticosteroids' use increase the risk of recurrence of pulmonary embolism).
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Krebs von den Lungen - 6 (KL-6) | 3 months
  a high molecular weight mucin-like glycoprotein expressed on cell surface of alveolar epithelial cells. Elevated levels of KL-6 occur in ILDs and it is recently widely accepted as a biomarker for diagnosis and prognosis of ILDs. Measured as (U/ml) using ELISA

SECONDARY OUTCOMES:
Respiratory Function Assessment; FEV1 | 3 months
  FEV1: Forced expiratory volume in the 1st second, measured in (% predicted) using a spirometer
Respiratory Function Assessment; FVC | 3 months
  FVC: Forced Vital Capacity which is the capacity of the lung to air volume, measured in (% predicted) using spirometer.
Respiratory Function Assessment; FEV/FVC Ratio | 3 months
  FEV/FVC: The ratio between the above 2 outcomes
Respiratory Function Assessment; 6MWD | 3 months
  6MWD: the distance walked by the patient after 6 minutes (measured in meters).
Respiratory Function Assessment; % O2 desaturation | 3 months
  % O2 desaturation: the amount of oxygen desaturation that occurs after walking for 6 minutes, measured as the difference between Spo2 before and after the patient walks for 6 minutes (% of oxygen saturation).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No